CLINICAL TRIAL: NCT07172464
Title: Early Feasibility Study (EFS) Evaluating Percutaneous Repair of the Atrial Septum With a Novel PFO Occluder: The PROTEA-PFO Study
Acronym: PROTEA-PFO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recross Cardio, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PL5001
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PFO; PFO - Patent Foramen Ovale; Cryptogenic Stroke; Patent Foramen Ovale; PFO-associated Stroke
Keywords: Patent Foramen Ovale; PFO; Cryptogenic Stroke; PFO Occluder; Transcatheter; PFO-associated stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Recross P3 Occluder (P3O) System (Experimental): The Recross P3 Occluder (P3O) is being developed for the purpose of transcatheter closure of a patent foramen ovale (PFO) to reduce the risk of recurrent ischemic stroke in patients with PFO-associated stroke.
  Interventions: Device: Recross P3 Occluder (P3O) System

INTERVENTIONS:
Device: Recross P3 Occluder (P3O) System — The Recross P3 Occluder (P3O) is being developed for the purpose of transcatheter closure of a patent foramen ovale (PFO) to reduce the risk of recurrent ischemic stroke in patients with PFO-associated stroke.

SUMMARY:
The goal of this clinical trial is to test a new heart device called P3 Occluder System in patients who have a small opening between the upper chambers of the heart (called a Patent Foramen Ovale or PFO) and have experienced a stroke that may be related to this heart opening. The main question it aims to answer is:

• Is the P3 Occluder System safe and effective for closing a PFO in patients who have had a stroke that could be related to a PFO.

Participants will:

* Undergo the procedure to implant the P3 Occluder System, if deemed appropriate.
* Visit their doctor at 1 month, 3 months, 6 months, 1 year, and 5 years after the procedure for follow up exams.
* Answer a phone call from study staff at 2 years, 3 years, and 4 years after the procedure to answer a survey.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 and ≤ 65 years of age
2. Diagnosis of PFO, defined as visualization of microbubbles per TEE in the left atrium within three cardiac cycles from the right atrial opacification demonstrating right-to-left shunting at rest and/or during Valsalva release.
3. Ischemic stroke, defined as acute focal neurological deficit, presumed to be due to focal ischemia and confirmed by MRI or CT to have a neuroanatomically relevant cerebral infarct.
4. Modified Rankin score (mRS) ≤ 3.
5. Appropriate PFO anatomy for implantation of the investigational device as evaluated and determined by independent committee.
6. Patient is willing and capable of providing informed consent.
7. Prior to index procedure (7-day window), persons of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

1. Other identifiable causes of stroke, including but not limited to aortic arch plaques (protruding >4 mm into the lumen), large artery atherosclerotic disease proximal to the territory of the index stroke, an established cardioembolic source, small-vessel occlusive disease, or arterial dissection, presence of left atrial appendage thrombus.
2. Other arteriopathy of the intracranial or extracranial vessels with >50% stenosis proximal to the territory of the index stroke.
3. Intracardiac thrombus or tumor.
4. Myocardial Infarction (MI) or unstable angina within the previous 180 days.
5. Life expectancy < 2 years.
6. Left ventricular aneurysm or akinesis.
7. Moderate to severe mitral valve stenosis or severe mitral regurgitation.
8. Aortic valve stenosis (mean gradient >20 mmHg) or severe regurgitation.
9. Active endocarditis or other infection that may preclude implantation of the investigational device.
10. Any valve vegetation or Lambl's excrescence of any left-sided valve.
11. Left ventricular dilated cardiomyopathy with LVEF <35%.
12. Another source of right-to-left shunts identified at baseline, including an atrial septal defect and/or fenestrated septum and pulmonary arteriovenous malformation.
13. History of atrial tachycardia, atrial fibrillation or flutter, AV block, or ventricular arrhythmia requiring antiarrhythmic medication, pacemaker, or AICD.
14. Severe renal failure ( Stage 4 CKD, eGFR <30) or patient requiring dialysis.
15. Severe liver disease (e.g., documented cirrhosis or active hepatitis).
16. Severe lung insufficiency (e.g., need for supplemental oxygen or chronic steroid medications).
17. Uncontrolled hypertension, defined as sustained elevated blood pressure >140/90 mm Hg.
18. Severe pulmonary artery hypertension, defined as pulmonary systolic pressure of >50mmHg.
19. Uncontrolled hyperglycemia, defined as HbA1c value >8% (IFCC: >64 mmol/mol).
20. Increased bleeding risk such as severe liver failure, active peptic ulcer, proliferative diabetic retinopathy, history of severe bleeding (e.g.: gastrointestinal bleeding, macroscopic hematuria, intraocular bleeding, intracranial or cerebral hemorrhage), or other history of bleeding or coagulopathy.
21. Known hypercoagulable state that would require full anticoagulation. Minimum testing to include lupus anticoagulant, anticardiolipin antibodies, beta-2-glycoprotein, homocysteine.
22. Subjects contraindicated for aspirin or clopidogrel.
23. Subjects not able to discontinue anticoagulation for indications other than then index stroke.
24. Any disorder in the investigator's opinion that could interfere with compliance of safety evaluation or require premature discontinuation of antiplatelet regime post-implantation, as well as any severe concurrent illness that would limit life expectancy (e.g., malignancies).
25. Currently an active subject in an investigational drug or device study that could confound the results of this study.
26. Any significant valve dysfunction that contraindicates PFO closure or increased pulmonary vascular resistance/severe pulmonary hypertension.
27. Contraindication for transesophageal echocardiography (TEE) or intracardiac echocardiography (ICE).
28. Any prior percutaneous cardiovascular intervention for AF ablation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Rate of Major Adverse Cardiovascular Events (MACE) | 30 days
  Rate of Major Adverse Cardiovascular Events (MACE) at 30 days post-procedure, defined as the composite of cardiac death (CD), myocardial infarction (MI), and stroke events.
Primary Performance Endpoint - Effective PFO Closure | 6 months
  Effective PFO Closure, at index procedure and at 6 months as measured by TEE, ad adjudicated.

SECONDARY OUTCOMES:
Secondary Safety Endpoints - Rate of device-related or procedure-related Serious Adverse Events (SAEs) | 30 days; 6 months
  Rate of device-related or procedure-related Serious Adverse Events (SAEs) at 30 days. Rate of device-related or procedure-related Serious Adverse Events (SAEs) at 6 months.
Secondary Performance Endpoint - Correct device position | 6 months
  Correct device position as assessed at 6 months on echocardiography, assessed by TTE or TEE.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York
  - Prisma Health - Upstate, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No